CLINICAL TRIAL: NCT02800616
Title: The Healthy Elementary School of the Future
Acronym: THESF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: UM MOVARE GGD
Record Dates: First submitted 2016-03-02; First posted 2016-06-15 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Overweight; Physical Activity; Malnutrition; Child Development; Lifestyle-related Condition; Socioeconomic Difficulty
Keywords: Academic Achievement; Accelerometry; Children; Primary school Intervention; Nutrition; Obesity; Physical Activity; Prevention; School Health
MeSH Terms: conditions — Overweight; Motor Activity; Malnutrition; Mental Disorders; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Full intervention group (Experimental): The full intervention ('The Healthy Primary School of the Future') is implemented in two schools involving extended school hours in which healthy nutrition, physical exercise, environmental, social, and educational activities are incorporated, during a period of four years.
  Interventions: Other: The Healthy Primary School of the Future
- Partial intervention group (Experimental): The partial intervention ('The Physical Activity School') is implemented in two other schools: involving extended school hours in which healthy nutrition, physical exercise, environmental, social, and educational activities are incorporated, during a period of four years. Hence, this intervention only differs from the full intervention on the absence of nutritional intervention. Instead, children bring their own food from home, as they normally do.
  Interventions: Behavioral: The Physical Activity School
- Control group (No Intervention): Four primary schools will function as control schools. The control schools have a representative Dutch school environment in terms of lifestyle education, school hours and amount of Physical Education (PE) lessons.

INTERVENTIONS:
Other: The Healthy Primary School of the Future — In two out of four intervention schools, a whole-school approach named 'The Healthy Primary School of the Future', is implemented with the aim of improving physical activity and dietary behaviour. For this intervention, pupils are offered an extended curriculum, including a healthy lunch, more physical exercises, and social and educational activities, next to the regular school curriculum.
  Arms: Full intervention group
Behavioral: The Physical Activity School — In the two other intervention schools, a physical-activity school approach called 'The Physical Activity School', is implemented, which is essentially similar to the other intervention, except that no lunch is provided.
  Arms: Partial intervention group

SUMMARY:
Unhealthy lifestyles in early childhood are a major global health challenge. These lifestyles often persist from generation to generation and contribute to a vicious cycle of health-related and social problems. We present a study protocol that examines the effectiveness of two novel, integrated healthy school interventions. One is a full intervention called 'The Healthy Primary School of the Future', the other is a partial intervention called 'The Physical Activity School'. These intervention approaches will be compared with the regular school approach that is currently common practice in the Netherlands. The main outcome measure will be changes in children's body mass index (BMI). In addition, lifestyle behaviours, academic achievement, child well-being, socio-economic differences, and societal costs will be examined.

DETAILED DESCRIPTION:
In close collaboration with various stakeholders, a quasi-experimental study was developed, for which children of four intervention schools (n = 1200) in the southern part of the Netherlands are compared with children of four control schools (n = 1200) in the same region. The interventions started in November 2015. In two of the four intervention schools, a whole-school approach named 'The Healthy Primary School of the Future', is implemented with the aim of improving physical activity and dietary behaviour. For this intervention, pupils are offered an extended curriculum, including a healthy lunch, more physical exercises, and social and educational activities, next to the regular school curriculum. In the two other intervention schools, a physical-activity school approach called 'The Physical Activity School', is implemented, which is essentially similar to the other intervention, except that no lunch is provided.

We hypothesize that these healthy school interventions will result in normalized BMI distributions that are more in line with national and international standards (smaller standard deviations) among primary school children, with a more pronounced effect in the full intervention schools (due to the expected synergy between exercise and diet) than in the partial intervention schools. Also, our multi-disciplinary research group will study a wide range of outcome measures, including lifestyle behaviours, academic achievement, child well-being, socio-economic differences, and societal costs. Moreover, an evaluation will be performed of the legal consequences of a healthy school approach in the Netherlands, as well as the conflicting interests of the stakeholders. Data collection is conducted within the school system. The interventions proceed during a period of four years. The baseline measurements started in September 2015 and yearly follow-up measurements are taking place until 2019.

Our primary research question is: What is the effect of the full intervention ('The Healthy Primary School of the Future') on the BMI of primary school children compared to no intervention (control schools)? Our secondary research question is: What is the effect of the full intervention on the BMI of primary school children compared to the partial intervention ('The Physical Activity School')? Our tertiary research questions are: (1) What is the effect of the full intervention in comparison with the partial intervention and the regular school approach (control schools) on: (a) children's levels of physical activity and sedentary behaviour, nutritional knowledge, healthy food preferences and behaviour, cognitive and non-cognitive performance, Health related-QoL, socio-emotional development, and sick leave? (b) parenting and teacher practices regarding physical activity and nutrition? (c) parental HR-QoL, well-being, labour participation and sick leave? (d) benefits across different socio-economic backgrounds? (e) long and short term cost-effectiveness? (f) satisfaction among the involved stakeholders (children, parents, teachers, and child care partners)? (2) Which determinants influence the quality of the implementation of the intervention? (3) What is the scope of children's human rights to health, what is the legal role of primary schools in realizing these rights (e.g., obligations and responsibilities of state and non-state actors, conflicts of interests and legal solutions to these conflicts), and is the intervention feasible within Dutch educational law?

A whole-school approach is a new concept in the Netherlands. Due to its innovative, multifaceted nature and sound scientific foundation, these integrated programmes have the potential to form a template for primary schools worldwide. The effects of this approach may extend further than the outcomes associated with well-being and academic achievement, potentially impacting legal and cultural aspects in our society.

ELIGIBILITY:
Inclusion Criteria:

* All children and their caregivers enrolled at one of the participating schools

Exclusion Criteria:

* None. Participants who switch schools during the four-year study period will not be followed-up.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2349 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Child absolute change in BMI Z-score, based on weight and height. | Four years
  Weight is measured using a weighing scale, to the nearest 0.1 kg; height is measured using a measuring rod, to the nearest 0.1 cm.

SECONDARY OUTCOMES:
Child hip and waist circumferences | Four years
  Using a measuring tape, to the nearest 0.1 cm, following the World Health Organization's assessment protocol
Child handgrip strength | Four years
  Measured using a calibrated Jamar hydraulic hand dynamometer to the nearest 0.5 kg
Child disease status | Four years
  Self-report measure (online parental questionnaire) since birth, hospital admissions (number and duration), healthcare visits (number), and medication use in the previous twelve months
Child pre-school blood pressure, birth weight, and information on disease history. | Obtained once
  Data previously obtained by the regional Public Health Services.
Parental BMI | Four years
  Self-report measure (online parental questionnaire).
Parental practices regarding nutrition | Four years
  Self-report measure (online parental questionnaire).Using the shortened version (nine items) of the Comprehensive Snack Parenting Questionnaire (CSPQ)
Parental practices regarding physical activity | Four Years
  Self-report measure (online parental questionnaire).questionnaire developed in the same style as he Comprehensive Snack Parenting Questionnaire (CSPQ)
Labour participation of parents | Four years
  Current employment status (self reported) is combined with parental education level and household income to determine socio economic status (SES).
Parents' ethnicity and level of (material) deprivation | Four years
  Self-report measure (online parental questionnaire).
Parental sick leave and absence from work or education because of illness of their child. | Four years
  Self-report measure (online parental questionnaire). Labour participation is combined with parental sick leave rates to determine productivity losses from work.
Child health-related quality of life | Four years
  Examined with the validated EuroQol 5-Dimensions Youth version questionnaire (EQ-5D-Y) and the proxy version for parents. Child-specific HR-QoL is measured by the validated Paediatric Quality of Life Inventory (PedsQL) and parents complete the proxy version of this questionnaire.
Child psychological attributes | Four years
  Assessed using the Strength and Difficulties Questionnaire.
Child social, emotional, and academic self-efficacy. | Four years
  Tested using the Self-Efficacy Questionnaire for Children (SEQ-C).
Child self-confidence, social skills, self-efficacy, school well-being, and social support | Four years
  Assessed with OnderwijsMonitor Limburg programme
Child physical activity and sedentary behavior (Actigraph accelerometer) | Four years
  In the week in which the child is wearing the accelerometer, parents fill in a short activity diary on their child's physical activity and swimming behaviour and exceptional circumstances (e.g., illness of the child)
Sports club membership, active forms of transport to school, and leisure time physical activities assessed in both children and parents. | Four years
  Self-report measure
Child food intake | Four years
  Assessed using a food frequency questionnaire and a dietary recall tool to be completed by both children and parents.
Child food preferences and familiarity with healthy food products. | Four years
  Self-report measure: The questions mainly consist of pictures of food items, for which children can indicate whether they have ever eaten these items and whether they like them or not.
Parental practices regarding nutrition and physical activity | Four years
  Self-report measure
Parental wellbeing | Four years
  measured by the Satisfaction With Life Survey (SWLS)
Parental health-related quality of life | Four years
  Measured with the EuroQol - 5-Dimensions Questionnaire (EQ-5D)
Socioeconomic status | Four years
  Self-report measure
School/ teacher practices regarding nutrition and physical activity | Four years
  E.g. modelling eating healthy food products and encouraging children's physical activity. Measured using adapted version of the Parental Practices Instrument
Teacher's self-reported height, weight and transport forms to work | Four years
  Written questionnaire
Child academic achievements | Four years
  Monitored using the Dutch national test called Centrale Eindtoets Basisonderwijs (CITO), and various other tests used by the schools. The CITO test measures language, maths and world orientation. In addition to the CITO test, many schools use a wide range of tests throughout the children's school careers. This also includes tests on maths (taken twice a year) and various aspects of language such as decoding skills, spelling, vocabulary, and reading comprehension.
School advice and the actual level of secondary school opted for (Dutch secondary education is hierarchically ordered). | Four years
  School registration system
School absenteeism and repeating classes | Four years
  School registration system
Process evaluation using a school satisfaction questionnaire | Four years
  Self-report measure: general parental satisfaction with their children's school (including safety, communication, quality of education, challenges to children, and professionalism of teachers). Implementation of the intervention is evaluated by qualitative outcome measures such as interviews with parents and children, and classroom observations.
Juridical evaluation through literature study and interviews | Four years
  Legal aspects will be addressed by a thorough scientific literature study and examination of policy and legislation instruments and case-law on the scope of children's right to health. Interviews with the parties involved in the healthy school setting will determine the juridical-related interests and possibilities.

CONTACTS AND LOCATIONS:
Overall Officials: Onno van Schayck, Prof. Dr., Principal Investigator — Professor at Maastricht University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hahnraths MTH, Willeboordse M, van Assema P, Winkens B, van Schayck CP. The Effects of the Healthy Primary School of the Future on Children's Fruit and Vegetable Preferences, Familiarity and Intake. Nutrients. 2021 Sep 17;13(9):3241. doi: 10.3390/nu13093241. PMID 34579117
- [Derived] Oosterhoff M, Jolani S, De Bruijn-Geraets D, van Giessen A, Bosma H, van Schayck OCP, Joore MA. BMI trajectories after primary school-based lifestyle intervention: Unravelling an uncertain future. A mixed methods study. Prev Med Rep. 2021 Jan 7;21:101314. doi: 10.1016/j.pmedr.2021.101314. eCollection 2021 Mar. PMID 33537184
- [Derived] Oosterhoff M, Over EAB, van Giessen A, Hoogenveen RT, Bosma H, van Schayck OCP, Joore MA. Lifetime cost-effectiveness and equity impacts of the Healthy Primary School of the Future initiative. BMC Public Health. 2020 Dec 9;20(1):1887. doi: 10.1186/s12889-020-09744-9. PMID 33297992
- [Derived] Oosterhoff M, van Schayck OCP, Bartelink NHM, Bosma H, Willeboordse M, Winkens B, Joore MA. The Short-Term Value of the "Healthy Primary School of the Future" Initiative: A Social Return on Investment Analysis. Front Public Health. 2020 Aug 21;8:401. doi: 10.3389/fpubh.2020.00401. eCollection 2020. PMID 32974255
- [Derived] Palacios Temprano J, Eichholtz P, Willeboordse M, Kok N. Indoor environmental quality and learning outcomes: protocol on large-scale sensor deployment in schools. BMJ Open. 2020 Mar 16;10(3):e031233. doi: 10.1136/bmjopen-2019-031233. PMID 32184302
- [Derived] Bartelink NHM, van Assema P, Kremers SPJ, Savelberg HHCM, Oosterhoff M, Willeboordse M, van Schayck OCP, Winkens B, Jansen MWJ. Can the Healthy Primary School of the Future offer perspective in the ongoing obesity epidemic in young children? A Dutch quasi-experimental study. BMJ Open. 2019 Oct 31;9(10):e030676. doi: 10.1136/bmjopen-2019-030676. PMID 31676651
- [Derived] Bartelink NHM, van Assema P, Jansen MWJ, Savelberg HHCM, Moore GF, Hawkins J, Kremers SPJ. Process evaluation of the healthy primary School of the Future: the key learning points. BMC Public Health. 2019 Jun 6;19(1):698. doi: 10.1186/s12889-019-6947-2. PMID 31170941
- [Derived] Boudewijns EA, Pepels JJS, van Kann D, Konings K, van Schayck CP, Willeboordse M. Non-response and external validity in a school-based quasi-experimental study 'The Healthy Primary School of the Future': A cross-sectional assessment. Prev Med Rep. 2019 Apr 17;14:100874. doi: 10.1016/j.pmedr.2019.100874. eCollection 2019 Jun. PMID 31061783
- [Derived] Oosterhoff M, Joore MA, Bartelink NHM, Winkens B, Schayck OCP, Bosma H. Longitudinal analysis of health disparities in childhood. Arch Dis Child. 2019 Aug;104(8):781-788. doi: 10.1136/archdischild-2018-316482. Epub 2019 Apr 4. PMID 30948361
- [Derived] Willeboordse M, Jansen MW, van den Heijkant SN, Simons A, Winkens B, de Groot RH, Bartelink N, Kremers SP, van Assema P, Savelberg HH, de Neubourg E, Borghans L, Schils T, Coppens KM, Dietvorst R, Ten Hoopen R, Coomans F, Klosse S, Conjaerts MH, Oosterhoff M, Joore MA, Ferreira I, Muris P, Bosma H, Toppenberg HL, van Schayck CP. The Healthy Primary School of the Future: study protocol of a quasi-experimental study. BMC Public Health. 2016 Jul 26;16:639. doi: 10.1186/s12889-016-3301-9. PMID 27456845
- See also: Official website about this project for various stakeholders (in Dutch) — http://www.degezondebasisschoolvandetoekomst.nl